CLINICAL TRIAL: NCT07252726
Title: A Randomised, Multicentre Trial Evaluating the Dose Timing (Morning vs Evening) of Endocrine-based Therapies in Metastatic Breast and Prostate Cancers (REaCT-CHRONO-MetBP Pilot Study)
Brief Title: Evaluating Dose Timing (Morning vs Evening) of Endocrine-based Therapies in Metastatic Breast and Prostate Cancers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-CHRONO-MetBP Pilot
Record Dates: First submitted 2025-09-18; First posted 2025-11-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Breast Cancer; Metastatic Prostate Cancer
Keywords: Chronotherapy; breast cancer; prostate cancer; endocrine therapy; metastatic cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: There will be 2 cohorts. Cohort A is for participants with breast cancer. Participants in Cohort A will be randomized to either morning or evening administration of endocrine-based therapy for breast cancer. Cohort B is for participants with prostate cancer. Participants in Cohort B will be randomized to either morning or evening administration of endocrine-based therapy for prostate cancer.
Masking Description: Participants and investigators will not be blinded to treatment allocation as the study is only randomizing treatment schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A, Arm A: Breast Cancer Cohort, Morning Group (Active Comparator): Participants with metastatic breast cancer in this arm are assigned morning administration of CDK4/6 inhibitor.
  Interventions: Other: Morning administration of CDK4/6 inhibitor
- Cohort A, Arm B: Breast Cancer Cohort, Evening Group (Active Comparator): Participants with metastatic breast cancer in this arm are assigned evening administration of CDK4/6 inhibitor.
  Interventions: Other: Evening administration of CDK4/6 inhibitor
- Cohort B, Arm A: Prostate Cancer Cohort, Morning Group (Active Comparator): Participants with metastatic prostate cancer in this arm are assigned morning administration of ARPI.
  Interventions: Other: Morning administration of ARPI
- Cohort B, Arm B: Prostate Cancer Cohort, Evening Group (Active Comparator): Participants with metastatic prostate cancer in this arm are assigned evening administration of ARPI.
  Interventions: Other: Evening administration of ARPI

INTERVENTIONS:
Other: Morning administration of CDK4/6 inhibitor — Morning administration of cyclin-dependent kinase (CDK) 4/6 inhibitor defined as, within one hour of the participant wake up time.
  Arms: Cohort A, Arm A: Breast Cancer Cohort, Morning Group
Other: Evening administration of CDK4/6 inhibitor — Evening administration of cyclin-dependent kinase (CDK) 4/6 inhibitor defined as, within one hour of the participant bedtime.
  Arms: Cohort A, Arm B: Breast Cancer Cohort, Evening Group
Other: Morning administration of ARPI — Morning administration of androgen receptor pathway inhibitors (ARPI) defined as, within one hour of the patient wake up time.
  Arms: Cohort B, Arm A: Prostate Cancer Cohort, Morning Group
Other: Evening administration of ARPI — Evening administration of androgen receptor pathway inhibitors (ARPI) defined as, within one hour of the patient bedtime.
  Arms: Cohort B, Arm B: Prostate Cancer Cohort, Evening Group

SUMMARY:
The REaCT-CHRONO-MetBP Pilot study will compare morning and evening administration of endocrine-based therapy in metastatic breast and prostate cancers.

Participants with metastatic breast or prostate cancer will be randomly placed in one of two groups: a morning group and an evening group. The group assignment will determine whether they take their endocrine therapy in the morning or the evening. The primary outcome of this pilot study is to evaluate the feasibility of study procedures in order to conduct a larger definitive trial in the future. The secondary outcomes include comparing quality of life, tolerability, and efficacy outcomes between the morning and evening groups for each of the two cancer cohorts (metastatic breast and prostate cancer).

ELIGIBILITY:
Cohort A (Breast Cohort) Inclusion Criteria

* Patients with metastatic hormonal receptor positive breast cancer
* Plan to receive endocrine therapy and a CDK4/6 inhibitor (either Ribociclib or Palbociclib) in the first-line metastatic setting
* Age ≥18 years
* Able to provide oral consent
* Willing and able to complete questionnaires as per study protocol

Cohort A (Breast Cohort) Exclusion Criteria

* Any contraindication in taking endocrine therapy and CDK4/6 inhibitor in the morning or evening
* Plan to receive abemaciclib (as this requires twice a day dosing)

Cohort B (Prostate Cancer) Inclusion Criteria

* Patients with metastatic castrate sensitive prostate cancer
* Plan to receive androgen receptor pathway inhibitor (either enzalutamide, apalutamide or abiraterone acetate) in combination with androgen deprivation therapy
* Age ≥18 years
* Able to provide oral consent
* Willing and able to complete questionnaires as per study protocol

Cohort B (Prostate Cancer) Exclusion Criteria

* Any contraindication in taking androgen receptor pathway inhibitor in the morning or evening
* Plan to receive darolutamide (as this requires twice a day dosing)
* Plan to receive docetaxel in combination with androgen receptor pathway inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility: accrual per site | 1 year
  Feasibility will be assessed according to a combination of metrics, including the accrual of at least 25 patients per cohort in one year for a total of three sites
Feasibility: participation rate | The accrual period, approximately 1 year
  Feasibility will be assessed according to a combination of metrics, including participation rate of at least 60% among patients approached.
Feasibility: number of participants who received allocated intervention | 4 weeks
  Feasibility will be assessed according to a combination of metrics, including at least 80% of enrolled patients receive treatment as per their allocated intervention for at least 4 weeks.

SECONDARY OUTCOMES:
Health-related quality of life: Functional Assessment of Cancer Therapy-General | Baseline and 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  Health-related quality of life using Functional Assessment of Cancer Therapy-General (FACT-G). Cohort A and Cohort B will answer the FACT-G. FACT-G has a score range of 0 to 108. Higher scores indicate better quality of life.
Health-related quality of life: Functional Assessment of Cancer Therapy-Endocrine Symptoms | Baseline and 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  Health-related quality of life using Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES). Cohort A and Cohort B will answer the FACT-ES. FACT-ES has a score range of 0 to 184. Higher scores indicate better quality of life.
Health-related quality of life: Functional Assessment of Cancer Therapy-Breast | Baseline and 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  Health-related quality of life using Functional Assessment of Cancer Therapy-Breast (FACT-B).
  Cohort A will complete the FACT-B. FACT-B has a score range of 0 to 148. Higher scores indicate better quality of life.
Health-related quality of life: Functional Assessment of Cancer Therapy-Prostate | Baseline and 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  Health-related quality of life using Functional Assessment of Cancer Therapy-Prostate (FACT-P).
  Cohort B will complete the FACT-P. FACT-P has a score range of 0 to 156. Higher scores indicate better quality of life.
Number of changes in treatment dose | 5 years
Number of treatment interruptions | 5 years
Number of treatment discontinuations | 5 years
Cohort A's adverse events of interest | 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  The number of participants in Cohort A that experience QTc prolongation, neutropenia, febrile neutropenia, hepatobiliary function.
Cohort B's adverse events of interest | 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  The number of participants in Cohort B that experience hypertension, hyperglycemia, rash, hypothyroidism, fatigue.
Adherence to treatment | 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  Adherence to treatment measured by the Five-Item Medication Adherence Report Scale (MARS-5 score). The MARS-5 has a range of 5-25. Higher scores indicate high adherence.
Participant preference in dose timing | Baseline
  Participants rank their preference on a scale of 0 to 10, where 0=prefer to take treatment in the morning, 5=no preference, 10=prefer to take treatment in the evening.

OTHER OUTCOMES:
Time to second-line systemic treatment | 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years
  Time from the randomization to start of second-line systematic treatment. This is reported on the Health Care Provider (HCP) follow up questionnaire which is completed at the various timepoints outlined in the time frame.
Overall survival | 4-, 12-, 26-, 52-weeks, 2-years, 3-years, 4-years, 5-years, 6-years post-randomization.
  Overall survival is the time from randomization to death from any cause. Survival status (yes/no) will be checked throughout the study at the various timepoints outlined in the time frame.
PSA reduction at 6 months | 6 months
  Cohort B only: prostate-specific antigen reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Savard, MD, Principal Investigator — The Ottawa Hospital; Ana-Alicia Beltran-Bless, MD, Principal Investigator — The Ottawa Hospital
Locations (3):
- Canada (3):
  - Waterloo Regional Health Network, Kitchener, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beltran-Bless AA, Vandermeer L, Ibrahim MFK, Hutton B, Shorr R, Savard MF, Clemons M. Does the Time of Day at Which Endocrine Therapy Is Taken Affect Breast Cancer Patient Outcomes? Curr Oncol. 2021 Jul 6;28(4):2523-2528. doi: 10.3390/curroncol28040229. PMID 34287262
- [Background] Savard MF, Ibrahim M, Saunders D, Pond GR, Ng TL, Awan AA, Sehdev S, Alqahtani N, Vandermeer L, MacDonald F, Beltran-Bless AA, Fallowfield L, Clemons M. A pragmatic, multicenter, randomized trial comparing morning versus evening dosing of adjuvant endocrine therapy (REaCT-CHRONO Study). NPJ Breast Cancer. 2025 May 29;11(1):49. doi: 10.1038/s41523-025-00762-7. PMID 40442096
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/